CLINICAL TRIAL: NCT06860126
Title: Design and Development of Strategies for Improving the Quality of Service and Utilization of Sporting and Recreational Places in the Municipality of Mashhad With the Approach to Elderly-Friendly City
Brief Title: Improving Sports and Recreation Services in Mashhad for Elderly and Intergenerational Interaction (ESPIRE-M)
Acronym: ESPIRE-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zinat Ebrahimi (Other)
Responsible Party: Sponsor-Investigator, Zinat Ebrahimi, Assistant Professor, Islamic Azad University, Sanandaj
Organization: Islamic Azad University, Sanandaj (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IR-IAU-MSHD.REC.1397.027
Record Dates: First submitted 2025-02-11; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Aged; Quality of Life; Mental Health
Keywords: Intergenerational Interaction; Age-Friendly City; Recreational Sports Facilities; Elderly Participation in Sports; Quality of Life in Seniors; Service Quality in Sports Facilities; SERVQUAL Questionnaire; SWOT Analysis for Elderly Sports; Yoga for Seniors; Light Aerobic Exercises for Elderly; Non-Sporting Intergenerational Programs; Health Outcomes in Elderly; Depression Reduction in Seniors; Social Engagement in Elderly; Mashhad Municipality Sports Programs; Elderly Well-Being; Urban Recreational Strategies; Inclusive Sports Programs; Physical Activity for Seniors; Psychological Health in Elderly
MeSH Terms: conditions — Psychological Well-Being | interventions — Yoga; Exercise; Control Groups

STUDY DESIGN:
Intervention Model Description: This study employs a Parallel Group interventional study model within a semi-experimental design framework. The methodology consists of two descriptive-correlational studies and a pre-test/post-test design with a control group.
  Research Design Participants were randomly assigned to six distinct groups: five experimental groups focused on different activities (intergenerational interaction, yoga exercises, exercise and interaction, park activities, and nursing home interaction) and one control group that maintained regular daily activities. This design allows for direct comparison of outcomes across groups and effectively assesses the interventions' relative effectiveness.
  Study Population and Sample Selection The study targeted elderly individuals aged 60 years and older, totaling 22,481, along with young participants aged 20 to 24 from Islamic Azad University. A cluster sampling method was employed to recruit 180 elderly participants, evenly divided by gender, along with 150 young
Who Masked: Participant, Outcomes Assessor
Masking Description: In addition to the roles specified above (Participant and Outcomes Assessor), the following parties are also masked in this clinical trial:
  1. Data Analysts: Individuals analyzing the trial data to prevent bias in the interpretation of results.
  2. Monitoring Entities: Independent monitors overseeing the trial, who are kept unaware of the treatment allocations to ensure objectivity in their assessments.
  This masking strategy helps maintain the integrity of the trial and reduces the risk of bias impacting the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental Group 1 (Experimental): * Tasks: Engage in 90-minute non-sport intergenerational interaction sessions, three times weekly for three months, in a controlled indoor environment. Activities include paired interactions and group discussions.
  * Participants: 60 seniors (30 women, 30 men) and 60 younger individuals (30 women, 30 men, average age 21.45 ± 0.35 years).
  Interventions: Behavioral: Intergenerational Activity Program: This indicates a program that involves activities designed for interaction between older adults and younger participants
- Experimental Group 2 (Experimental): * Tasks: Participate in 90-minute intergenerational yoga sessions, three times weekly for three months, in a gym setting. Sessions include warm-up, yoga exercises (asanas and pranayama), and relaxation.
  * Participants: 60 seniors (30 women, 30 men) and 60 younger individuals (30 women, 30 men).
  Interventions: Behavioral: Yoga and Mindfulness Sessions
- Experimental Group 3 (Experimental): * Tasks: Engage in 60-minute light aerobic exercises in a park, followed by 30-minute group discussions, three times weekly for three months.
  * Participants: 60 seniors (30 women, 30 men) and 60 younger individuals (30 women, 30 men).
  Interventions: Behavioral: Physical Exercise and Storytelling
- Experimental Group 4 (Experimental): * Tasks: Participate in 90-minute non-exercise intergenerational interaction sessions in a park, focusing on group discussions and storytelling.
  * Participants: 60 seniors (30 women, 30 men) and 60 younger individuals (30 women, 30 men).
  Interventions: Behavioral: Outdoor Interaction Games
- Experimental Group 5 (Experimental): * Tasks: Engage in 90-minute non-exercise intergenerational interaction sessions in a nursing home, focusing on group discussions and storytelling.
  * Participants: 60 seniors (30 women, 30 men) and 60 younger individuals (30 women, 30 men).
  Interventions: Behavioral: Social Visits to Nursing Homes
- Control Group (Other): * Tasks: Continue daily routines without intergenerational interaction or structured activities.
  * Participants: 78 seniors (39 women, 39 men) selected through stratified random sampling.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: Intergenerational Activity Program: This indicates a program that involves activities designed for interaction between older adults and younger participants — Engage in 90-minute intergenerational interaction sessions, three times a week for three months, in a controlled indoor environment.
  * Spend the first 45 minutes actively interacting with a younger participant in pairs, collaborating on activities of interest to the senior.
  * Participate in group activities such as book reading, puzzles, joke-telling, and sharing experiences for the remaining 45 minutes.
  * Attend 36 sessions held on odd days in the main hall of the Neshat Center.
  * Gender Representation:
  * 60 participants (30 women and 30 men) aged 60 and above, selected through stratified random sampling from Mashhad's elderly population.
  * 60 younger participants (30 women and 30 men) with an average age of 21.45 ± 0.35 years, selected through purposive sampling from Mashhad's Islamic Azad University.
  Arms: Experimental Group 1
Behavioral: Yoga and Mindfulness Sessions — Participate in 90-minute intergenerational yoga sessions, three times a week for three months, in a gym setting.
  * Perform modified yoga exercises suitable for seniors, including:
  * 20 minutes of warm-up with stretching and joint rotations.
  * 50 minutes of main exercises (asanas and pranayama).
  * 20 minutes of relaxation and meditation (Shavasana).
  * Attend sessions on odd days at 9 AM in the Neshat Center yoga hall.
  * Gender Representation:
  * 60 participants (30 women and 30 men) aged 60 and above, selected through stratified random sampling from Mashhad's elderly population.
  * 60 younger participants (30 women and 30 men) with an average age of 21.45 ± 0.35 years, selected through purposive sampling from Mashhad's Islamic Azad University.
  Arms: Experimental Group 2
Behavioral: Physical Exercise and Storytelling — Engage in 60-minute light aerobic exercises, three times a week for three months, in a park setting.
  * Follow warm-up and aerobic exercises led by a senior fitness instructor.
  * Spend 30 minutes in a friendly group discussion, sharing experiences and memories with younger participants.
  * Attend sessions on even days at 9 AM in Mashhad's Mellat Park.
  * Gender Representation:
  * 60 participants (30 women and 30 men) aged 60 and above, selected through stratified random sampling from Mashhad's elderly population.
  * 60 younger participants (30 women and 30 men) with an average age of 21.45 ± 0.35 years, selected through purposive sampling from Mashhad's Islamic Azad University.
  Arms: Experimental Group 3
Behavioral: Outdoor Interaction Games — Participate in 90-minute intergenerational interaction sessions, three times a week for three months, in a park setting.
  * Engage in non-exercise activities such as group discussions, storytelling, and sharing experiences with younger participants.
  * Attend sessions on even days at 9 AM in Mashhad's Mellat Park.
  * Gender Representation:
  * 60 participants (30 women and 30 men) aged 60 and above, selected through stratified random sampling from Mashhad's elderly population.
  * 60 younger participants (30 women and 30 men) with an average age of 21.45 ± 0.35 years, selected through purposive sampling from Mashhad's Islamic Azad University.
  Arms: Experimental Group 4
Behavioral: Social Visits to Nursing Homes — Engage in 90-minute intergenerational interaction sessions, three times a week for three months, in a nursing home setting.
  * Participate in non-exercise activities such as group discussions, storytelling, and sharing experiences with younger participants.
  * Attend sessions on odd days at 9 AM in the nursing home.
  * Gender Representation:
  * 60 participants (30 women and 30 men) aged 60 and above, selected through stratified random sampling from Mashhad's elderly population.
  * 60 younger participants (30 women and 30 men) with an average age of 21.45 ± 0.35 years, selected through purposive sampling from Mashhad's Islamic Azad University.
  Arms: Experimental Group 5
Other: control group — Continue with their daily routines without participating in any intergenerational interaction or structured activities.
  * No specific interventions or programs are provided.
  * Gender Representation:
  * 78 participants (39 women and 39 men) aged 60 and above, selected through stratified random sampling from Mashhad's elderly population.
  Arms: Control Group

SUMMARY:
This interventional study aims to design strategies to improve service quality and productivity in recreational sports facilities in Mashhad Municipality, focusing on creating an age-friendly city. The research consists of two parts: fieldwork and an experimental section.

Field Section:

1. Assess seniors' perceptions of services using the SERVQUAL questionnaire and other tools.
2. Conduct a SWOT analysis to identify strengths, weaknesses, opportunities, and threats related to elderly sports participation.

Experimental Section:

Evaluate the impact of intergenerational sports activities on elderly participants (aged 60+). Participants were paired with younger individuals and randomly allocated to five groups, including a control group.

Group Tasks:

* Control Group: 78 seniors continued daily routines without structured activities.
* Experimental Groups:

  1. Non-sport intergenerational interaction sessions (90 minutes, 3x/week).
  2. Intergenerational yoga sessions (90 minutes, 3x/week).
  3. Light aerobic exercises + group discussions (90 minutes, 3x/week).
  4. Non-exercise intergenerational sessions in a park (90 minutes, 3x/week).
  5. Non-exercise intergenerational sessions in a nursing home (90 minutes, 3x/week).

     Field Study Sample:
* 384 customers of Mashhad Municipality sports facilities (192 women, 192 men).

Key Notes:

* Elderly participants were selected through cluster sampling; younger participants were purposively sampled from Mashhad's Islamic Azad University.
* Gender balance (50% women, 50% men) was maintained in all groups.

Main Questions:

1. How do service quality factors influence customers of Mashhad Municipality sports facilities?
2. Do intergenerational programs improve quality of life, health, and well-being for seniors?
3. What are the strengths, weaknesses, opportunities, and threats for elderly sports participation?
4. What strategies can enhance elderly participation in sports?

DETAILED DESCRIPTION:
1. Data Collection Instruments

The following questionnaires will be utilized to achieve the research objectives:

1. Demographic Characteristics Questionnaire: Includes variables such as age, gender, marital status, income, education level, occupation, and number of children.
2. Socio-economic Status Questionnaire: Assesses various dimensions of socio-economic status.
3. World Health Organization Quality of Life Questionnaire: Measures quality of life based on established criteria.
4. Elderly Depression Questionnaire: Assesses depression levels among elderly participants.
5. General Health Questionnaire (GHQ-28): A self-administered tool examining overall health, focusing on non-psychotic disorders.
6. Parent-Child Relationship Scale: Evaluates the dynamics of relationships between parents and their children.
7. Student Depression Questionnaire: Measures depression levels among university students.
8. Service Quality Questionnaire: Assesses the quality of services provided.
9. Facility Checklist and Productivity Index Checklist: Tools for evaluating facility conditions and efficiency.
10. World Health Organization Age-Friendly City Criteria Questionnaire: Assesses compliance with age-friendly city standards.

2. Study Population and Sample Selection

The study population includes two groups:

* Elderly Participants: Individuals aged 60 years and older residing in Mashhad. Recruitment will occur through public announcements and notices in locations such as parks and mosques, aiming to enroll 150 elderly individuals using purposive and convenient sampling.
* Young Participants: Students aged 20 to 24 years enrolled at Islamic Azad University. A total of 100 students (50 male, 50 female) will be recruited through public announcements and notices posted in all faculties during the academic year 2017-2018.

After collecting demographic data and completing questionnaires, elderly participants will be randomly assigned to three groups: two experimental groups and one control group. The sample size is based on experimental research designs, with a larger number selected to enhance generalizability and reduce dropout rates.

3. Limitations of the Study

* Lack of accurate data on the number of active elderly individuals and their participation levels in regular sports activities.
* Cultural barriers limiting women's participation in community activities.
* Limited access to organizations specializing in elderly issues, restricting the ability to obtain a representative sample.

  4. Ethical Considerations
* Participants will be informed about the study's objectives and methodology before participation.
* Informed consent will be obtained from all participants.
* Confidentiality of personal information will be maintained.
* Private interpretations of results will be offered to interested individuals.
* No financial burden will be imposed on participants.
* The study will comply with religious and cultural standards relevant to participants and the broader community.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Elderly Participants:

Aged 60 years or older.

Ability to engage in physical activities.

Absence of sensory or motor disabilities.

No use of antidepressant medications.

No history of conditions such as Alzheimer's or other illnesses that could pose risks during exercise.

Younger Participants:

Aged 20 to 24 years.

Unmarried.

Living with their parents.

Native residents of Mashhad.

Exclusion Criteria:

Irregular attendance (more than two absences).

Physical or psychological issues hindering participation.

Lack of willingness to continue.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is open to all self-identified genders. Participants aged 60 years and older will be recruited equally from all gender identities, ensuring inclusivity and representation. For the young participants aged 20 to 24 years from Islamic Azad University, both male and female individuals, regardless of gender identity, are eligible to participate.
Enrollment: 384 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Effects of Intergenerational Interventions on Quality of Life Effects of Intergenerational Interventions on Quality of Life Effects of Intergenerational Interventions on Quality of Life | Baseline and after a 3-month intervention period.
  Quality of Life (QOL) was assessed using the World Health Organization Quality of Life Questionnaire (Short Form), a 26-item tool measuring four dimensions: physical health, psychological health, social relationships, and environment. Items are rated on a 6-point scale, with scores converted to a 0-100 scale. Higher scores indicate better QOL.
  * Pre-Test Scores:
    * Physical Health: Range = 12.5-68.75
    * Psychological: Range = 31.25-62.5
    * Social Relationships: Range = 37.5-50
    * Environment: Range = 25-62.5
  * Post-Test Scores:
    * Physical Health: Range = 25-68.75
    * Psychological: Range = 18.75-62.5
    * Social Relationships: Range = 28.125-46.875
    * Environment: Range = 12.5-37.5
  * Results:
    * Physical health: 41.53 (baseline) → 70.97 (post-intervention).
    * Psychological: 40.93 → 63.31.
    * Social relationships: 42.94 → 50.20.
    * Environment: 44.15 → 52.62.
Effects of Intergenerational Interventions on Mental Health (General Health) | Baseline and after a 3-month intervention period.
  Mental health was assessed using the General Health Questionnaire (GHQ-28), a 28-item tool evaluating physical symptoms, anxiety, social functioning, and depression. Items are scored from 0 to 3, with total scores ranging from 0-84. Higher scores indicate greater psychological distress.
  Pre-test Scores:
  Somatic symptoms: 4-21
  Anxiety and sleep disorder: 2-21
  Social function: 7-21
  Depression symptoms: 9-21
  Total: 29-70
  Post-test Scores:
  Somatic symptoms: 5-21
  Anxiety and sleep disorder: 1-21
  Social function: 7-20
  Depression symptoms: 7-21
  Total: 30-68
  * Somatic symptoms: 13.61 (baseline) → 8.78 (post-intervention).
  * Anxiety and sleep disorder: 13.62 → 7.27.
  * Social function: 15.48 → 11.95.
  * Depression symptoms: 13.57 → 6.63.
Effects of Intergenerational Interventions on Depression Levels | Measurements were taken at baseline and after a 3-month intervention period.
  Depression levels were measured using the Geriatric Depression Scale (Short Form), a 15-item binary response questionnaire specifically designed for the elderly. Scores range from 0-15, with higher scores indicating greater depression.
  Pre-test Scores: 8-15
  Post-test Scores: 5-14

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Zinat Ebrahimi, Professor, Principal Investigator — Physical Education and Sport, Islamic Azad Sanandaj, Iran.
Locations (2):
- Iran (2):
  - Department of Physical Education and Sport Science, Islamic Azad University, Sanandaj, Iran., Sanandaj, Kurdistan Province
  - Department of Physical Education and Sport Science, Faculty of Humanities and Literature, Sanandaj Branch, Islamic Azad University, Sanandaj, Iran., Sanandaj, Kurdistan Province

IPD SHARING:
Plan to Share IPD: No
Due to persistent technical difficulties in providing a functional web address for the IPD sharing plan on the clinical trial site, interested parties are encouraged to contact zin368@gmail.com for further information. We have encountered issues that prevent the proper display or access of the sharing link, necessitating this alternative means of communication.

REFERENCES:
- [Background] Ebrahimi, Zinat. Helen Nazary, Parivash Piraki. (2023). The Service Quality of Sport-entertainment Facilities of Mashhad Municipality with the Approach of an Elderly-friendly City in 2018 (Persian). Journal of Gerontology (joge), 7(4): 89-100. DOI: 10.22034/JOGE.7.4.8. https://joge.ir/article-1-618-fa.html
- [Background] Veisi, K. Ismailzadeh Ghandehary, M.R. Ebrahimi, Z. (2023). Comparing the Effectiveness of Interventions of Intergenerational Interaction and Physical Activities on Depression of Elderly Women and Men (Persian). Journal of Gerontology (joge). 8(1): 10-19. https://joge.ir/article-1-620-fa.html
- [Background] Ebrahimi Z, Esmaeilzadeh Ghandehary MR, Veisi K. Comparing the efficacy of Yoga exercise and intergenerational interaction program on mental health of elderly. J Research & Health2019; 9(5): 401- 410.
- [Background] Eshun-Wilson I, Siegfried N, Akena DH, Stein DJ, Obuku EA, Joska JA. Antidepressants for depression in adults with HIV infection. Cochrane Database Syst Rev. 2018 Jan 22;1(1):CD008525. doi: 10.1002/14651858.CD008525.pub3. PMID 29355886
- [Background] Steptoe A, Deaton A, Stone AA. Subjective wellbeing, health, and ageing. Lancet. 2015 Feb 14;385(9968):640-648. doi: 10.1016/S0140-6736(13)61489-0. Epub 2014 Nov 6. PMID 25468152
- [Background] Santini S, Tombolesi V, Baschiera B, Lamura G. Intergenerational Programs Involving Adolescents, Institutionalized Elderly, and Older Volunteers: Results from a Pilot Research-Action in Italy. Biomed Res Int. 2018 Dec 5;2018:4360305. doi: 10.1155/2018/4360305. eCollection 2018. PMID 30627555
- [Background] Murayama Y, Ohba H, Yasunaga M, Nonaka K, Takeuchi R, Nishi M, Sakuma N, Uchida H, Shinkai S, Fujiwara Y. The effect of intergenerational programs on the mental health of elderly adults. Aging Ment Health. 2015;19(4):306-14. doi: 10.1080/13607863.2014.933309. Epub 2014 Jul 10. PMID 25010219
- [Background] Murayama Y, Murayama H, Hasebe M, Yamaguchi J, Fujiwara Y. The impact of intergenerational programs on social capital in Japan: a randomized population-based cross-sectional study. BMC Public Health. 2019 Feb 6;19(1):156. doi: 10.1186/s12889-019-6480-3. PMID 30727981
- [Background] Mosor E, Waldherr K, Kjeken I, Omara M, Ritschl V, Pinter-Theiss V, Smolen J, Hubel U, Stamm T. An intergenerational program based on psycho-motor activity promotes well-being and interaction between preschool children and older adults: results of a process and outcome evaluation study in Austria. BMC Public Health. 2019 Mar 1;19(1):254. doi: 10.1186/s12889-019-6572-0. PMID 30823911
- [Background] Luanaigh CO, Lawlor BA. Loneliness and the health of older people. Int J Geriatr Psychiatry. 2008 Dec;23(12):1213-21. doi: 10.1002/gps.2054. PMID 18537197
- [Background] Kamei T, Itoi W, Kajii F, Kawakami C, Hasegawa M, Sugimoto T. Six month outcomes of an innovative weekly intergenerational day program with older adults and school-aged children in a Japanese urban community. Jpn J Nurs Sci. 2011 Jun;8(1):95-107. doi: 10.1111/j.1742-7924.2010.00164.x. Epub 2010 Dec 9. PMID 21615702
- [Background] Halpin SN, Dillard RL, Idler E, Clevenger C, Rothschild E, Blanton S, Wilson J, Flacker JM. The benefits of being a senior mentor: Cultivating resilience through the mentorship of health professions students. Gerontol Geriatr Educ. 2017 Jul-Sep;38(3):283-294. doi: 10.1080/02701960.2015.1079707. Epub 2015 Aug 7. PMID 26251869
- [Background] Di Martino G, Della Valle C, Centorbi M, Buonsenso A, Fiorilli G, Crova C, di Cagno A, Calcagno G, Iuliano E. Bridging Generations Through Movement: "How and Why" Intergenerational Programs Operate-A Systematic and Narrative Review. Geriatrics (Basel). 2024 Oct 22;9(6):139. doi: 10.3390/geriatrics9060139. PMID 39449376
- [Background] Bruce ML. Psychosocial risk factors for depressive disorders in late life. Biol Psychiatry. 2002 Aug 1;52(3):175-84. doi: 10.1016/s0006-3223(02)01410-5. PMID 12182924
- [Background] Barbosa, M. R., Campinho, A., & Silva, G. (2021). "give and receive": The impact of an intergenerational program on institutionalized children and older adults. Journal of Intergenerational Relationships, 19(3), 283-304.
- [Background] Au, A., Ng, E., Garner, B., Lai, S., & Chan, K. (2015). Proactive aging and intergenerational mentoring program to promote the well-being of older adults: pilot studies. Clinical Gerontologist, 38(3), 203-210.
- [Background] Alonso-Cortes Fradejas B, Lafuente-Ureta R, Calvo S, Fernandez-Gorgojo M, Poveda-Lopez JL, Jimenez-Sanchez C. Analysis of an intergenerational service-learning experience based on physical exercise in a community setting: a mixed-method study. Front Public Health. 2025 Jan 14;12:1509016. doi: 10.3389/fpubh.2024.1509016. eCollection 2024. PMID 39926288